CLINICAL TRIAL: NCT07126171
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Clinical Study on the Efficacy and Safety of Reduning Injection in the Treatment of Chikungunya Fever
Brief Title: A Clinical Study on the Efficacy and Safety of Reduning Injection in the Treatment of Chikungunya Fever
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYZY-RDN-Ⅴ-CHIKF-202504
Record Dates: First submitted 2025-08-04; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chikungunya Fever
MeSH Terms: conditions — Chikungunya Fever | interventions — reduning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduning treatment group (Experimental): Redunign Injection, intravenous drip, 20 ml per dose, once a day
  Interventions: Drug: Reduning injection
- placebo group (Placebo Comparator): The simulant of Reduning Injection, for intravenous drip, 20 ml per time, once a day
  Interventions: Drug: The simulant of Reduning Injection

INTERVENTIONS:
Drug: Reduning injection — reduning Injection, intravenous drip, 20 ml per time, once a day;
  Arms: Reduning treatment group
Drug: The simulant of Reduning Injection — The simulant of Reduning Injection, for intravenous drip, 20 ml per time, once a day
  Arms: placebo group

SUMMARY:
To evaluate the efficacy and safety of Reduning Injection in the treatment of chikungunya fever

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter clinical study of the efficacy and safety of Reduning Injection in the treatment of Chikungunya fever. The purpose of this study is to evaluate the efficacy and safety of Reduning Injection in the treatment of Chikungunya fever. The study uses the IWRS system to randomize the study participants, adopts the double-blind method, selects placebo control, plans to be conducted simultaneously in multiple research centers across the country, plans to include 400 study participants, and randomly assigns them to the test drug group and the placebo group at a 1:1 ratio, with 200 participants in the test drug group.

ELIGIBILITY:
Inclusion criteria:

1. Meet the diagnostic criteria for chikungunya fever (can be randomly selected based on suspected cases);
2. Fever duration ≤ 48 hours, and at the time of consultation, axillary temperature ≥ 38.0℃ (if antipyretic drugs have been taken, the axillary temperature must be ≥ 38.0℃ 4 hours or later after taking the drugs);
3. The first symptoms of chikungunya fever other than fever have a duration ≤ 72 hours;
4. At the time of consultation, have one or more of the following symptoms: headache, back pain or generalized muscle pain, nausea and vomiting, joint pain, joint swelling, joint stiffness, rash, and the severity is moderate or above;
5. Age between 18 and 70 years old (including both ends), gender not restricted;
6. Provide informed consent and sign the informed consent form.

Exclusion criteria:

1. Those diagnosed with dengue fever, alphavirus infection, influenza, novel coronavirus infection, infectious erythema, post-infection arthritis (including rheumatic fever), scarlet fever, rickettsial diseases (typhus, scrub typhus), measles, drug-induced rash, etc.;
2. Acute, chronic stages of chikungunya fever and high-risk populations;
3. Those with severe primary diseases of the cardiovascular, liver, kidney and hematopoietic systems;
4. Those with chronic arthritis;
5. Those with immunodeficiency (such as AIDS patients, those with long-term use of corticosteroids or other immunosuppressive drugs resulting in weakened immune function);
6. Those with obesity (BMI ≥ 30 kg/m2) or weight < 40 kg;
7. Those suspected or confirmed to have alcohol addiction, drug abuse history, or those with cognitive impairment, severe mental illness and unable to cooperate with the clinical study;
8. Pregnant women or those preparing for pregnancy within 6 months, and lactating women;
9. Those with allergic constitution, such as history of allergy to two or more drugs or foods, or those known to be allergic to the drugs used in this study and the ingredients of acetaminophen tablets;
10. Those who participated in any clinical study within 3 months before the screening examination;
11. Those judged by the researcher to be not suitable to participate in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2025-11-26 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Duration of symptoms | -1 day to 0 day, medication duration of 5 days ± 1 day, onset of disease 14 days ± 2 days after the onset, 90 days ± 3 days after the onset
  The time from the first administration of the medication until all scores for the symptoms of chikungunya fever were 0 or 1 points (if the score was 1 before the medication, it must be reduced to 0), and this remained stable for 48 hours or more

SECONDARY OUTCOMES:
Recovery time of body temperature | The subjects recorded these information in the "Subject Diary Card" during the period from -1 day to 0 day, 5 days ± 1 day after medication administration, and 14 days ± 2 days after the onset of the disease.
  The time required for the axillary temperature to be ≤ 37.0℃ after medication administration and to remain at this level for 24 hours or more
Time for fever reduction to take effect | The subjects recorded these information in the "Subject Diary Card" during the period from -1 day to 0 day, 5 days ± 1 day after medication administration, and 14 days ± 2 days after the onset of the disease.
  The time required for the first drop of 0.5℃ or more in axillary temperature after medication administration
The change in the integer VAS score for joint pain from baseline after 5 days of medication and 14 days after the onset of the disease | After taking the medicine for 5 days, 14 days after the onset of the disease
  The severity of joint pain was evaluated using the Visual Analogue Scale (VAS). This method employed a 100mm long straight line, where 0 represented no joint pain symptoms and 100 represented the most intense pain. The research participants marked the corresponding position on the line that indicated their most severe level of pain. This was recorded during visits 1 to 3 in the "Research Participant Diary Card". The recording points were as follows: The first time, record the most severe pain level within 0.5 hours before the first medication administration; thereafter, record the most severe pain level once at 08:00 and 20:00 each day, with a time window of ±1 hour; if the score is 0 for more than 48 hours, there is no need to record again.
The change in the number of joint pain episodes compared to the baseline value | The researchers conducted evaluations on the study participants once each at -1 day to 0 day, 5 days ± 1 day after medication administration, and 14 days ± 2 days after the onset of the disease.
Time for disappearance of individual symptoms | -1 day to 0 day, medication duration of 5 days ± 1 day, onset of disease 14 days ± 2 days after the onset, 90 days ± 3 days after the onset
  The symptom score after medication administration was 0, and the duration required for it to remain at this score for 24 hours or longer.
The rate of disappearance of individual symptoms | -1 day to 0 day, medication duration of 5 days ± 1 day, onset of disease 14 days ± 2 days after the onset, 90 days ± 3 days after the onset
  The symptom score after medication administration was 0, and the duration required for it to remain at this score for 24 hours or longer.
The incidence rate of complications (such as bleeding, hematoma, encephalitis, myelitis, etc.) | From -1 day to 0 day, and up to 90 days ± 3 days after the onset of the disease, the occurrence of complications by the subjects will be recorded by the researchers.
  The incidence rate of complications (such as bleeding, hematoma, encephalitis, myelitis, etc.)
The usage situation of emergency medications | From -1 day to 0 day, within 5 days ± 1 day after medication administration, and 14 days ± 2 days after the onset of the disease.
  The subjects should record in the "Subject Diary Card" before each use of emergency medication.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China